CLINICAL TRIAL: NCT06464484
Title: The Effects Of Probiotics On Stress And Bowel Habits Among Healthy Adults From Umm Al-Qura University at Makkah: A Randomized Interventional Study
Brief Title: The Effects Of Probiotics On Stress Among Healthy Adults From Umm Al-Qura University At Makkah
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Essra Noorwali, Associate Professor, Umm Al-Qura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-2023-01-1414
Record Dates: First submitted 2024-06-12; First posted 2024-06-18 (Actual); Last update posted 2024-06-20 (Actual); Status verified 2024-06

CONDITIONS: Stress; Constipation; Anthropometry; Bowel Disease
Keywords: Probiotics; Saudi Arabia; Stress; Gut-brain axis; Gastrointestinal tract
MeSH Terms: conditions — Constipation; Intestinal Diseases | interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: This intervention was a randomized, controlled trial. The participants were randomized using lottery method either to the probiotic group (PG) and the control group (CG). The probiotic group received a daily (Lactobacillus rhamnosus GG 6x10^9 cpu) supplement for 30 days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: cases (Experimental): Consumed one probiotic for 30 days everyday with or without food. Dicoflor 60 probiotic supplements were provided that contained Lactobacillus rhamnosus GG (ATCC 53103) that contained 6x10^9 colony forming units (cpu)) per capsule.
  Interventions: Dietary Supplement: Probiotics (Lactobacillus rhamnosus GG (ATCC 53103)
- Controls (No Intervention): Had high stress levels but did not consume probiotics

INTERVENTIONS:
Dietary Supplement: Probiotics (Lactobacillus rhamnosus GG (ATCC 53103) — Already mentioned in arm/group descriptions
  Other Names: Dicoflor 60
  Arms: Experimental: cases

SUMMARY:
The goal of this clinical trial is to study the effects of probiotic supplementation on stress levels and bowel habits in healthy Saudi adults for both males and females.

The main questions it aims to answer are:

Does probiotic supplementation decrease stress levels? Does probiotic supplementation improve bowel habits?

Researchers compared between the intervention group receiving probiotic supplements with high stress levels with a control group not receiving probiotics with high stress levels to see if probiotics decreases stress levels.

DETAILED DESCRIPTION:
Participants were required to

1. Attend a visit to the nutrition clinic at Umm AL-Qura University to assess for eligibility.
2. Eligible participants were asked to sign a consent form and anthropometrics, stress, bowel habits, food records and knowledge on probiotics were collected
3. Participants were randomized based on lottery based method to an interventional or control group
4. Intervention group received 30 capsules of probiotics (Lactobacillus rhamnosus GG, 6x10^9 cpu) to be taken once daily
5. After 30 days, all participants had to attend a second visit at the nutrition clinic at Umm Al-Qura University to assess stress levels, bowel habits and receive their incentives (discount voucher of restaurants).

ELIGIBILITY:
Inclusion Criteria:

* Students at Umm Al-Qura University
* Age ≥ 18 years
* Healthy individuals
* Both genders
* Saudi nationality

Exclusion Criteria:

* Diagnosed with chronic illness or/and psychiatric condition
* Consumption of medications or supplements in the previous 3 months
* Pregnant and breastfeeding
* Smoker

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 85 (Actual)
Dates: Start 2023-01-26 (Actual); Primary Completion 2024-03-31 (Actual); Study Completion 2024-04-30 (Actual)

PRIMARY OUTCOMES:
Stress | Post intervention at 30 days
  Perceived stress scale (PSS) was used in both English and Arabic versionsndividual scores on the PSS can range from 0 to 40 with higher scores indicating higher perceived stress.
  Scores ranging from 0-13 would be considered low stress. Scores ranging from 14-26 would be considered moderate stress. Scores ranging from 27-40 would be considered high perceived stress.
Bowel function | Post intervention at 30 days
  The questionnaire was developed to collect, comorbid illnesses, a prescription list, and specific questions related to bowel habits including fluid intake, usual diet, fecal matter consistency, frequency of defecation, and straining. The questionnaire also contained questions about laxative usage, previous surgeries, and lifestyle. The questionnaire was translated by an authorised translator and was based on a previous study.

CONTACTS AND LOCATIONS:
Overall Officials: Essra Noorwali, PhD, Principal Investigator — Umm Al-Qura University
Locations (1):
- Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
The following may be shared:
  Study Protocol Statistical Analysis Plan (SAP) Informed Consent Form (ICF) Clinical Study Report (CSR) Analytic Code

REFERENCES:
- [Derived] Noorwali EA, Aljaadi AM, Abusudah WF, Bakhdar FA, Bin-Ali DH, Alshinawi A, Bawazir A, Mutlaq RA, Maimany HA, Barnawi LA, Murshed B, Aljared B, Azzeh FS. The effect of probiotic supplementation on perceived stress and bowel function in healthy young adults: evidence from a randomized controlled trial in Makkah. Front Nutr. 2026 Jan 6;12:1717047. doi: 10.3389/fnut.2025.1717047. eCollection 2025. PMID 41567324